CLINICAL TRIAL: NCT04109365
Title: Electrical Epidural Stimulation Test for Confirmation of Epidural Catheter Placement in Labouring Women
Brief Title: Obstetric Placement Study Using EST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Chi-Ho Ban Tsui, Professor-Med Ctr Line, Stanford University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 52856
Record Dates: First submitted 2019-09-11; First posted 2019-09-30 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Obstetric Pain; Anesthesia, Local
Keywords: Electrical Epidural Stimulation Test
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Electrical Epidural Stimulation Test (EST) (Experimental): Laboring women are given EST test initially before local anesthetic is administered and 1 hour post-anesthetic in order to measure sensory and motor responses.
  Interventions: Diagnostic Test: Electrical Epidural Stimulation Test (EST)

INTERVENTIONS:
Diagnostic Test: Electrical Epidural Stimulation Test (EST) — EST measures sensory/motor responses

SUMMARY:
Combined spinal-epidural (CSE) is an established technique for providing labour analgesia to obstetric patients which provides rapid onset but unsustained analgesia. The epidural catheter can be used to extend and provide continuous pain relief, however during single-segment needle-through-needle CSE, the catheter is untested. This study aims to confirm placement of epidural catheters of anesthesia through the epidural stimulation test (EST) which was first described by the PI of the study for confirming placement of epidural catheters approximately 20 years ago.

ELIGIBILITY:
Inclusion Criteria:

* Females, 18 years and older
* American Society of Anesthesiologists physical status I or II
* Full-term pregnancy with request for epidural early in labour (i.e. Regular labor or C-Section)

Exclusion Criteria:

* Contraindication to regional anesthesia
* Allergy or hypersensitivity to lidocaine, bupivacaine, or fentanyl
* Use of sedatives or opioids
* Abnormal vertebrae anatomy
* Neurological disorder with lumbar involvement
* Implanted electronic devices

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Obstetric related study
Enrollment: 40 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Electrical Epidural Stimulation Test | Duration of EST test (approximately 1-2 hours)
  Investigate the ability of the electrical epidural stimulation test (EST) to determine the position of the epidural catheter anesthesia for labour analgesia after low-dose anesthetic as compared to the gold standard of clinical assessment.

SECONDARY OUTCOMES:
Pain Scores | Approximately 3 hours following introduction of anesthetics through the catheter.
  Patients will be asked for a pain score by research staff approximately 3 hours following placement of the epidural catheter and low-dose anesthetics are introduced. The pain scores will be on a scale from 0-10 with 0 representing no pain and 10 representing maximum pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Lucille Packard Children's Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Carvalho JC, Khemka R, Loke J, Tsui BC. Low-dose intrathecal local anesthetic does not increase the threshold current for the epidural stimulation test: a prospective observational trial of neuraxial analgesia in labouring women. Can J Anaesth. 2015 Mar;62(3):265-70. doi: 10.1007/s12630-014-0291-x. Epub 2014 Dec 11. PMID 25501494